CLINICAL TRIAL: NCT04391816
Title: COVID-19 Pandemic Impact on Alcohol (PIA) - A Natural History Study
Status: Recruiting | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200115; 20-AA-0115
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10-09

CONDITIONS: Alcohol Drinking; Alcohol-Related Disorders; Pandemic; Psychological Stress
Keywords: Coronavirus; Alcohol Use Disorder; SARS-CoV2; Stress; Social Isolation; Natural History
MeSH Terms: conditions — Alcohol Drinking; Alcohol-Related Disorders; Stress, Psychological; Coronavirus Infections; Alcoholism; Social Isolation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Participants that were previously enrolled in the NIAAA Screening Protocol.

SUMMARY:
Background:

The SARS-CoV-2 virus has caused a pandemic infection called COVID-19. It is a global threat to people, communities, and health systems. Researchers are concerned about the mental health effects of the pandemic. They want to learn more about how it is affecting people s alcohol use and problems, and how it may continue to affect them over time.

Objective:

To study the impact of the COVID-19 pandemic on alcohol use and consequences in individuals across the spectrum of alcohol use and those with alcohol use disorder.

Eligibility:

Participants who have been screened under the NIAAA Screening, Assessment and Management Protocol (14-AA-0181)

Design:

Participants will complete a baseline survey by phone. It will ask about alcohol use, alcohol dependence, and stress. It covers 2 time periods: the 12 months before the pandemic started and the time since it started.

Participants will get an ID code and a link to an online survey. They will complete the online survey within a week of the phone survey.

Participants will complete a series of online surveys over 24 months. For the first year, surveys will be completed weekly for the first 4 weeks, then biweekly for the next 8 weeks, and then every 1-2 months for the rest of the year. For the second year, surveys will be completed every 6 months. Surveys will cover the following topics:

* Alcohol use and its consequences
* Other substance use
* Stress
* Impact of the COVID-19 pandemic
* Pain
* Physical health
* Sleep
* Quality of life.

Because the course of the pandemic may change, the frequency of the surveys may change.

Participation lasts 2 years.

DETAILED DESCRIPTION:
Study Description:

The novel coronavirus (SARS-CoV-2) outbreak started in 2019 and has resulted in a world-wide pandemic infection designated COVID-19. This pandemic has become an unprecedented global threat to individuals, communities and health systems. While immediate attention has appropriately focused on prevention and treatment of SARS CoV-2 infection, the widespread societal mental health consequences of the pandemic cannot be ignored. Given the catastrophic impact of the COVID-19 pandemic, it is critical to prospectively and longitudinally assess the impact on alcohol use and problems, along with associated behaviors and outcomes. Thus, the goal of this study is to examine the impact of the COVID-19 pandemic on alcohol use and consequences in individuals across the spectrum of alcohol use and alcohol use disorder.

Objectives:

The specific aims of this study are:

1. To evaluate the impact of the COVID-19 pandemic on alcohol consumption and consequences in individuals across the spectrum of alcohol use and those with AUD.
2. To evaluate the time-course of changes in measures of negative life events, social isolation and stress, and their effect on alcohol consumption and consequences over a 2-3 year period during and following the COVID-19 pandemic.
3. (Exploratory aim) To examine the role of anxiety, depression, craving, binge drinking, impaired control in the relationships examined above.

Endpoints:

In Phase 1 of the study (conducted from June 2020-September 2023), participants will be invited to complete several surveys by phone and/or online over 2 years at intervals that range from weekly to bimonthly in the first year and every 6 months during the second year. Depending on the trajectory of the pandemic, the frequency of the surveys may be modified if necessary. In Phase 2 of the study (starting in October 2023), participants will complete surveys by phone and/or online over 3 years at 1 to 3-month intervals. The surveys will assess a range of outcomes related to alcohol consumption and consequences, along with measures of other substance use, stress, sleep, physical health and quality of life.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Participants who have enrolled in the NIAAA Natural History Protocol (14-AA-0181) and completed screening and phenotyping assessments.
2. Willing and able to complete frequent (weekly to monthly) surveys either online or by phone.

EXCLUSION CRITERIA:

As this is a natural history protocol, there are no formal exclusionary criteria for this study. Participants who are determined by the interviewer to be uncooperative or unable to provide consent via telephone will not be enrolled into the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population for this study includes healthy adults across the spectrum of alcohol use who have been screened under the NIAAA screening protocol (14-AA-0181). This sample includes non-drinkers, light drinkers, non-treatment-seeking heavy drinkers, and treatment-seeking individuals with alcohol use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AUDIT Score | 24 months
  Alcohol Use Disorder Identification Test (AUDIT): This is a 10-item questionnaire designed to screen for AUD. The first 3 questions constitute the AUDIT-C and provides a measure of alcohol consumption. The total score provides a continuous quantification of AUD severity.
ADS Score | 24 months
  Alcohol Dependence Scale (ADS): This 25-item scale will be used to measure severity of alcohol dependence. This scale covers alcohol withdrawal symptoms, impaired control over drinking, awareness of a compulsion to drink, increased tolerance to alcohol, and salience of drink-seeking behavior.

SECONDARY OUTCOMES:
Life Events Questionnaire (LEQ) Score | 24 monhts
  Life Events Questionnaire (LEQ): This questionnaire assesses positive and negative life events and their impact on participants
UCLA Loneliness Scale (UCLA-LS) Score | 24 months
  UCLA Loneliness Scale (UCLA-LS): This is a 20-item scale designed to measure a person s subjective feeling of loneliness and social isolation in the last month
Perceived Stress Scale (PSS) Score | 24 months
  Perceived stress scale (PSS): This is a 10-item scale to measure perception of stress

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- NIAAA Section on Human Psychopharmacology, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerda M, Tracy M, Galea S. A prospective population based study of changes in alcohol use and binge drinking after a mass traumatic event. Drug Alcohol Depend. 2011 May 1;115(1-2):1-8. doi: 10.1016/j.drugalcdep.2010.09.011. Epub 2010 Oct 24. PMID 20977977
- [Background] Druss BG. Addressing the COVID-19 Pandemic in Populations With Serious Mental Illness. JAMA Psychiatry. 2020 Sep 1;77(9):891-892. doi: 10.1001/jamapsychiatry.2020.0894. No abstract available. PMID 32242888
- [Background] Clay JM, Parker MO. Alcohol use and misuse during the COVID-19 pandemic: a potential public health crisis? Lancet Public Health. 2020 May;5(5):e259. doi: 10.1016/S2468-2667(20)30088-8. Epub 2020 Apr 8. No abstract available. PMID 32277874
- [Derived] Agarwal K, Luk JW, Stangl BL, Schwandt ML, Momenan R, Goldman D, Diazgranados N, Kareken DA, Leggio L, Ramchandani VA, Joseph PV. Parosmia Is Positively Associated With Problematic Drinking, as Is Phantosmia With Depressive Symptoms. J Addict Med. 2024 Sep-Oct 01;18(5):567-573. doi: 10.1097/ADM.0000000000001332. Epub 2024 May 22. PMID 38776446
- [Derived] Luk JW, Stangl BL, Gunawan T, Schwandt ML, Morris JK, Axelowitz JC, Chawla S, Lee BA, Carraco M, Walsh S, McDuffie C, Agarwal K, Joseph PV, Momenan R, Goldman D, Diazgranados N, Ramchandani VA. Changes in Alcohol-Related Behaviors and Quality of Life During the COVID-19 Pandemic: Impact of Alcohol Use Disorder Diagnosis and Treatment History. J Clin Psychiatry. 2022 Nov 7;84(1):22br14462. doi: 10.4088/JCP.22br14462. No abstract available. PMID 36350598
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-AA-0115.html